CLINICAL TRIAL: NCT00601120
Title: Pilot Feasibility Protocol of RF Ablation of Treatment of Metastatic Lesions in Patients Undergoing Antiangiogenic Therapy for Stage IV Renal Cell Carcinoma
Brief Title: RF Ablation of Treatment of Metastatic Lesions in Patients Undergoing Antiangiogenic Therapy for Stage IV Renal Cell Carcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This protocol was never officially opened and no patients were recruited.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Rupal Bhatt, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-287
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Renal Cell Carcinoma
Keywords: antiangiogenic therapy; RF ablation
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Needles are inserted into the tumor(s) under guidance by a CT scan or ultrasound. The electrodes in the needles will be heated up to 202 degrees Fahrenheit and will remain heated for up to 12 minutes.
  Other Names: RF Ablation

SUMMARY:
The purpose of this study is to look at the effects of a procedure called radiofrequency ablation on kidney tumors from patients who are undergoing antiangiogenic treatment. Antiangiogenic treatment is a type of treatment that inhibits formation of new blood vessels that are required for tumor growth. Radiofrequency ablation (RF ablation) involves inserting a needle into tumor tissue and administering heat to the tumor tissue that is sufficient to kill the tumor cells.

DETAILED DESCRIPTION:
* Participants will undergo a RF ablation procedure of one or more of their tumors that have not gone away while they have been undergoing antiangiogenic treatment. The RF ablation procedure will be performed in the operating room at one of the Dana-Farber/Harvard Cancer Center hospitals and will be performed under general anesthesia.
* Blood will also be drawn 2-4 weeks before the procedure, at the time of teh procedure and 2-4 weeks after the procedure.
* The RF ablation procedure will be performed at specified times in relation to the participants antiangiogenic treatment (sorafenib or sunitinib): a) If the participant is taking sorafenib, they will be asked to stop taking it 2-5 days prior to the RF ablation procedure; b) if the participant is taking sunitinib, they will be asked to stop taking it 4-7 days prior to the RF ablation procedure.
* Participants will have an MRI or a CT scan of their tumor(s) within 2-4 weeks of the procedure and 2-4 weeks after the procedure. The MRI or CT will scan the tumor(s) to determine how much blood flow is going to them.
* At the time of RF ablation, participants will have a biopsy of their tumor(s) and will receive a CT scan in the area the ablation was performed after the procedure to assess for any bleeding. They will also be monitored for 4 hours after the RF ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are on antiangiogenic therapy for a minimum of 4 weeks and have isolated metastatic lesions showing either persistence or resistance to therapy that might benefit from local therapy such as RF ablation.
* Male or female patients 18 years of age or older
* Clinical, radiographic, or pathologic diagnosis of clear cell RCC
* Ongoing treatment with sorafenib or sunitinib, off clinical trials
* Acceptable risk for general anesthesia in the judgement of the study investigator and by the department of anesthesiology upon preoperative testing.
* At least one lesion that has not completely resolved while on antiangiogenic therapy
* Candidate lesions of 1cm or greater in diameter
* Safe access to the tumor for a needle placed under ultrasound guidance
* ECOG Performance Status of 0 or 1
* Adequate bone marrow, and renal as assessed by the laboratory requirements outlined in the protocol

Exclusion Criteria:

* History of bleeding diathesis or unexpected surgical bleeding
* Patients currently on anticoagulation
* Medical contraindication to MR imaging (pacemaker, metal debris in eye, etc.)
* Prior RF to the index tumor
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety, toxicity and feasibility of RFA for the treatment of metastatic lesion in patients undergoing antiangiogenic therapy. | 3 years

SECONDARY OUTCOMES:
To evaluate the efficacy of RF ablation by measurement of diameter of ablation for treatment in this patient population. | 3 years
To evaluate relative efficacy of RFA in treatment of metastatic lesions showing sensitivity vs. resistance to anti-angiogenic therapy. | 3 years
To examine the mechanism of resistance to antiangiogenic therapy by examining the pathologic findings in sensitive and resistant metastatic lesions in patients with RCC treated with sorafenib and sunitinib. | 3 years
To study the relationship of peripheral blood angiogenic markers and vascular imaging to molecular changes within the tumor in sensitive and resistant metastatic lesions. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rupal Bhatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States